CLINICAL TRIAL: NCT06473259
Title: Evaluation of Clinical Outcomes of Chemotherapy or Androgen-receptor Targeting Therapy (Alone or in Combination) or Radiotherapy on the Primary Tumor in Combination With Androgen Deprivation Therapy in Metastatic Hormone-sensitive Prostate Cancer: Multicenter Observational Study of Patients Undergoing Treatment in Clinical Practice in Italian Hospitals
Brief Title: Evaluation of Clinical Outcomes of Chemotherapy or Androgen-receptor Targeting Agent (Alone or Combined) or Radiotherapy on Primary Tumor in Addition to Androgen Deprivation Therapy in HOrmone-Sensitive Metastatic Prostate Cancer Patients
Acronym: ECHOS
Status: Recruiting | Type: Observational
Sponsor: Santa Chiara Hospital (Other)
Responsible Party: Principal Investigator, Orazio Caffo, Director, Santa Chiara Hospital
Other Study IDs: A349
Record Dates: First submitted 2024-05-28; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer; Hormone Sensitive Prostate Cancer; Metastatic Tumor
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Docetaxel; apalutamide; enzalutamide; Abiraterone Acetate; darolutamide; Radiotherapy; Triptorelin Pamoate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ADT + docetaxel: mHSPC patients treated with ADT + docetaxel
  Interventions: Drug: Docetaxel; Drug: Triptorelin
- ADT + ARPI: mHSPC patients treated with ADT + ARPI
  Interventions: Drug: Apalutamide Oral Tablet; Drug: Enzalutamide Oral Tablet; Drug: Abiraterone acetate tablets; Drug: Triptorelin
- ADT + ARPI + docetaxel: mHSPC patients treated with ADT + docetaxel + ARPI
  Interventions: Drug: Docetaxel; Drug: Darolutamide Oral Tablet; Drug: Triptorelin
- ADT + radiotherapy on primary tumor: mHSPC patients treated with ADT + radiotherapy on primary tumor
  Interventions: Radiation: radiotherapy; Drug: Triptorelin

INTERVENTIONS:
Drug: Docetaxel — 6 courses of docetaxel 75 mg/sqm iv
  Groups: ADT + ARPI + docetaxel; ADT + docetaxel
Drug: Apalutamide Oral Tablet — 240 mg /daily orally
  Groups: ADT + ARPI
Drug: Enzalutamide Oral Tablet — 600 mg /daily orally
  Groups: ADT + ARPI
Drug: Abiraterone acetate tablets — 1000 mg /daily orally
  Groups: ADT + ARPI
Drug: Darolutamide Oral Tablet — 600 mg/daily orally
  Groups: ADT + ARPI + docetaxel
Radiation: radiotherapy — radical radiotherapy on primary tumor
  Groups: ADT + radiotherapy on primary tumor
Drug: Triptorelin — 3,75 mg im/4 w

SUMMARY:
The aim of this observational study is to evaluate the clinical outcomes of treatment with docetaxel, ARTA (alone or in combination) or with radiotherapy on the primary tumor for mCSPC, in an unselected population, in clinical practice

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed diagnosis of adenocarcinoma of the prostate, metastatic, not undergoing previous treatment (except hormone therapy initiated no more than 4-6 months prior to docetaxel) for metastatic disease
2. treatment with docetaxel, ARPI (alone or in combination) or with radiation therapy on the primary tumor in combination with ADT within normal clinical practice or expanded access programs initiated between January 2015 and December 2027.
3. availability of inpatient and/or outpatient medical records for clinical data collection

Exclusion Criteria:

1. histological diagnosis other than adenocarcinoma
2. patients who have received multiple lines of ADT for mCSPC
3. patients who have received docetaxel or ARTA for metastatic castration-resistant disease

Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: All patients with mCSPC who initiated treatment with docetaxel, ARPI (alone or in combination) or with radiotherapy on the primary tumor in addition to ADT within clinical practice or expanded access programs in Italian hospitals from January 2015 to December 2027 will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-12-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | From date of treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  the projected rate over the time of patients without progressive disease

SECONDARY OUTCOMES:
overall survival | From date of treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  the projected rate over the time of alive patients

OTHER OUTCOMES:
rate of patients with an objective response | through study completion, an average of 2 year
  rate of patients who experienced a reduction of at least 30% of measurable lesions

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Azienda Ospedaliera San Luigi, Orbassano, Torino
  - Istituto Oncologico Veneto, Padua
  - Santa Chiara Hospital, Trento

IPD SHARING:
Plan to Share IPD: Undecided